CLINICAL TRIAL: NCT04413656
Title: cfDNA Methylation Assay for Clinical Evaluation of Patients With Stage IA Lung Cancer After Ablation Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Chief Physician, Department of Pulmonary Medicine, Director, Department of Respiratory Endoscopy and Interventional Pulmonology, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCHE201902
Record Dates: First submitted 2019-11-11; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2019-06

CONDITIONS: Lung Cancer
Keywords: ablation; circulating free DNA; methylation
MeSH Terms: conditions — Lung Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ablation group (Experimental): Patients with stage IA inoperable peripheral lung tumor will be performed ablation. cfDNA methylation would be monitored at different times(before surgery , after surgery 1month, 3month, and every 3month in the first year and every 6 months in the second ). Meanwhile, post-treatment response will be evaluated and follow up will be carried out according to the standard procedure.
  Interventions: Other: ablation
- surgery group (Experimental): Patients with stage IA operable peripheral lung tumor will be performed surgery. cfDNA methylation would be monitored at different time(before surgery , after surgery 1month, 3month). Post-treatment response will be evaluated and follow up will be carried out according to the standard procedure.
  Interventions: Other: surgery

INTERVENTIONS:
Other: ablation — Patients with stage IA inoperable peripheral lung tumor will be performed ablation. cfDNA methylation would be monitored at different times(before surgery , after surgery 1month, 3month, and every 3month in the first year and every 6 months in the second ).
  Arms: ablation group
Other: surgery — Patients with stage IA inoperable peripheral lung tumor will be performed ablation. cfDNA methylation would be monitored at different times(before surgery, after surgery 1month, 3month).
  Arms: surgery group

SUMMARY:
The objective is to screen and monitor the efficacy of cfDNA methylation in patients with stage I lung cancer after ablation, to compare the similarities and differences of cfDNA methylation between surgical treatment and ablation in patients with stage I lung cancer, and to look for new indicators to assess the efficacy of ablation therapy and to monitor lung cancer recurrence.

DETAILED DESCRIPTION:
The objective is to screen and monitor the efficacy of cfDNA methylation in patients with stage I lung cancer after ablation, to compare the similarities and differences of cfDNA methylation between surgical treatment and ablation in patients with stage I lung cancer, and to look for new indicators to assess the efficacy of ablation therapy and to monitor lung cancer recurrence.

The main research content is to screen the cfDNA methylation index that can monitor the efficacy of stage I lung cancer ablation and compare the similarities and differences of cfDNA methylation in patients with stage I lung cancer after surgery and ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-85 years old;
2. The peripheral pulmonary nodules found in patients with chest CT, preoperative examination showed that the clinical stage of patients was T1N0M0, IA;
3. patients are not suitable for surgical treatment through multidisciplinary assessment, agree to accept ablation
4. Patients have good compliance with the tests and follow-ups, understand the situation of the study and sign informed consent.

Exclusion Criteria:

1. The patient is generally in poor condition and cannot tolerate the examination;
2. patients with a cardiac pacemaker or stent in the heart; peripheral tumors of the lungs are adjacent to large blood vessels or important structures;
3. patients with poor compliance;
4. Researchers believe that it is not appropriate to participate in this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-12-17 (Estimated); Study Completion 2021-06-17 (Estimated)

PRIMARY OUTCOMES:
Screening and monitoring the change of cfDNA methylation index | before surgery , after surgery 1month, 3month, 6month，9month，12month，18month and 24month
  Screening and monitoring the change of cfDNA methylation index in patients with stage I lung cancer after ablation

SECONDARY OUTCOMES:
Comparing similarities and differences between cfDNA methylation in surgical treatment and ablation | before surgery , after surgery 1month, 3month
  Comparing similarities and differences between cfDNA methylation in surgical treatment and ablation of patients with stage I lung cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No